CLINICAL TRIAL: NCT02377180
Title: Capsaicin-induced Muscle Pain in Humans: From Investigating Central Pain Processing to Developing Clinical Applications
Brief Title: Capsaicin-induced Muscle Pain in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 066/13
Record Dates: First submitted 2015-02-11; First posted 2015-03-03 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
Keywords: musculoskeletal pain; regional anesthesia; diagnostic nerve block; intramuscular capsaicin; referred pain; hyperalgesia; experimental pain; central hypersensitivity; human experimental pain
MeSH Terms: conditions — Musculoskeletal Pain; Pain, Referred; Hyperalgesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 (Experimental): Intramuscular injection of capsaicin for the study of pain and hyperalgesia
  Interventions: Procedure: Intramuscular capsaicin injection
- Part 2 (Active Comparator): Pain arising from supraspinatus muscle vs. pain arising from trapezius muscle. Nerve block is only expected to be effective in the former.
  Interventions: Procedure: Suprascapular nerve block
- Part 3 (Active Comparator): Suprascapular nerve block vs. intramuscular local anesthetic against pain arising from the supraspinatus muscle.
  Interventions: Procedure: Local anesthetic infiltration

INTERVENTIONS:
Procedure: Intramuscular capsaicin injection — Intramuscular injection of capsaicin: 50 mcg/0.5 ml
  Arms: Part 1
Procedure: Suprascapular nerve block — Injection of capsaicin 50 mcg/0.5 ml into the supraspinatus or trapezius muscle in randomized order, followed by suprascapular nerve block (ultrasound-guided) using Lidocaine 1%; nerve block is expected to be effective only in pain arising from the supraspinatus muscle. Trapezius pain serves as control condition.
  Evaluates the diagnostic validity of suprascapular nerve block for muscle pain.
  Arms: Part 2
Procedure: Local anesthetic infiltration — Injection of capsaicin 50 mcg/0.5 ml into the supraspinatus muscle in two different sessions; suprascapular nerve block in one session and intramuscular local anesthetic infiltration in one session (in randomized order) using Lidocaine 1%; the aim is to investigate which procedure provides faster and more efficient pain relief. Compares effectivity of suprascapular nerve block vs. intramuscular local anesthetic infiltration.
  Arms: Part 3

SUMMARY:
There is currently no specific diagnostic test for primary muscular pain. The present study investigates whether selective blockade of the suprascapular nerve can effectively abolish experimental pain arising from the supraspinatus muscle. Experimental muscle pain is induced by intramuscular injection of capsaicin, an alkaloid from red chili peppers. The study consists of three parts:

1. to describe the development, time course and intensity of capsaicin-induced muscle pain
2. to evaluate the effectiveness of suprascapular nerve block against capsaicin-induced muscle pain
3. to compare suprascapular nerve block and direct intramuscular local anesthetic infiltration for their effectiveness in capsaicin-induced muscle pain

DETAILED DESCRIPTION:
Background

Musculoskeletal pain is one of the most common reasons for consulting a physician. Many musculoskeletal pain disorders are associated with a widespread decrease in pain thresholds, indicating a state of hyperexcitability of the central nervous system.

This central hypersensitivity can be assessed by measuring pain thresholds to different experimental stimuli, using so-called quantitative sensory tests (QST).

Several experimental pain models are being used in healthy volunteers in order to study the central mechanisms of pain processing. Injection of capsaicin is one of them, which is associated with spreading of local pain, development of referred pain and hyperalgesia to thermal, mechanical or electrical stimuli.

Intramuscular injection of capsaicin is therefore potentially interesting for investigating primary muscle pain, central hypersensitivity and endogenous pain modulation. The present research project comprises three substudies which use intramuscular capsaicin to detect changes in central pain processing and to evaluate clinical tools for the diagnosis of primary muscle pain.

Part 1: The investigators hypothesize that the intensity, duration and expansion area of capsaicin-induced muscle pain depends on a subject's endogenous pain modulation. The investigators expect that subjects with strong endogenous pain modulation develop less pain and hyperalgesia after capsaicin injection than subjects with poor endogenous pain modulation. A large sample of healthy volunteers will therefore be screened using QST and then recruited for capsaicin injection if they show either very strong or very weak endogenous pain modulation. The data of the whole sample can be used to determine normative values of endogenous pain modulation.

Part 2 investigates the ability of suprascapular nerve block to abolish primary muscle pain. Healthy volunteers will receive capsaicin injection into the supraspinatus muscle or the trapezius muscle as a control condition in a randomized, blinded fashion. The investigators expect that the nerve block is more effective in the former compared to the latter muscle.

Part 3 compares the analgesic efficacy of suprascapular nerve block and direct intramuscular local anesthetic infiltration of the supraspinatus muscle after capsaicin injection. This will determine which procedure is more effective to treat primary muscle pain.

Objective

1. To determine normative values for endogenous pain modulation in healthy volunteers
2. To demonstrate that capsaicin-induced pain and hyperalgesia depend on endogenous pain modulation
3. To calculate sensitivity and specificity of suprascapular nerve block for the diagnosis of primary muscle pain
4. To determine whether suprascapular nerve block or intramuscular local anesthetic infiltration are more effective against muscle pain

Methods

1. intramuscular injection of capsaicin
2. quantitative sensory tests (pressure pain thresholds)
3. ultrasound-guided suprascapular nerve block
4. ultrasound-guided intramuscular local anesthetic infiltration

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Written informed consent

Exclusion Criteria

* Any acute pain at the moment of testing
* Intake of analgesics 24hours before testing
* Intake of antidepressants, anticonvulsants or benzodiazepines
* Allergy to local anesthetic or skin disinfectant
* Pregnancy or breast-feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Intensity of shoulder pain on numeric rating scale | two hours

SECONDARY OUTCOMES:
Pressure pain thresholds | two hours
Area of referred pain | two hours

CONTACTS AND LOCATIONS:
Overall Officials: Michele Curatolo, M.D., Ph.D., Study Chair — Department of Anesthesiology and Pain Therapy, University of Washington, Seattle WA, USA
Locations (1):
- University Department of Anesthesiology and Pain Therapy,Inselspital Bern, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] Graven-Nielsen T, Gibson SJ, Laursen RJ, Svensson P, Arendt-Nielsen L. Opioid-insensitive hypoalgesia to mechanical stimuli at sites ipsilateral and contralateral to experimental muscle pain in human volunteers. Exp Brain Res. 2002 Sep;146(2):213-22. doi: 10.1007/s00221-002-1169-7. Epub 2002 Jul 13. PMID 12195523
- [Background] Witting N, Svensson P, Gottrup H, Arendt-Nielsen L, Jensen TS. Intramuscular and intradermal injection of capsaicin: a comparison of local and referred pain. Pain. 2000 Feb;84(2-3):407-12. doi: 10.1016/s0304-3959(99)00231-6. PMID 10666547
- [Background] Siegenthaler A, Moriggl B, Mlekusch S, Schliessbach J, Haug M, Curatolo M, Eichenberger U. Ultrasound-guided suprascapular nerve block, description of a novel supraclavicular approach. Reg Anesth Pain Med. 2012 May-Jun;37(3):325-8. doi: 10.1097/AAP.0b013e3182409168. PMID 22222688